CLINICAL TRIAL: NCT00540852
Title: Monitoring the Response of Chemotherapy on Breast Cancer Tumor by Photon Migration Spectroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other); Chao Family Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, David Hsiang, M.D., Division of Surgical Oncology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Purpose: Device Feasibility
Other Study IDs: 20022306
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer receiving chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic Tool (Other): Diffuse Optical Spectroscopy Imaging
  Interventions: Device: Diffuse Optical Spectroscopy Imaging

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy Imaging — Diffuse Optical Spectroscopy Imaging

SUMMARY:
Optimal management of patients with locally advanced breast cancer remains a complex therapeutic problem. Newly diagnosed breast cancers in the United States with a higher incidence in medically underserved areas. The optimal intensity and duration of neoadjuvant chemotherapy still remains controversial due to the difficulty of evaluating response to therapy. The goal would be to prevent over and under treatment of patients with neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The Researcher developed a diagnostic device called Diffuse Optical Spectroscopy Imaging is a non-invasive optical technique that utilizes intensity-modulated, near-infrared light to quantitatively measure optical properties in thick tissues.

Diffuse Optical Spectroscopy Imaging can images tissue hemoglobin , oxygen saturation, blood volume fraction, water content, fat content and cellular structure. The measurements provide quantitative optical property values that reflect changes in tissue perfusion, oxygen consumption, and cell/matrix development.

There is no therapeutic benefit to the subject, especially none that might influence the indication for the diagnostic procedure as indicated. However, information obtained may lead to a new form of non-invasive imaging for the early detection of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female non-pregnant and age greater than or equal to 21 years old but less than 75 years old
* Diagnosed with breast cancer and will be receiving neoadjuvant chemotherapy

Exclusion Criteria:

* Female pregnant and age less than 21 years old and have no diagnosis of breast cancer

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2002-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic tool | 12 weeks
  Diffuse Optical Spectroscopy Imaging Breast Cancer Tumor in the response of Chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: David Hsiang, M.D, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (2):
- United States (2):
  - Beckman Laser Institute University Of California Irvine, Irvine, California
  - Chao Family Comprehensive Cancer Center, Orange, California